CLINICAL TRIAL: NCT00126659
Title: A Phase II Neoadjuvant Clinical Trial to Evaluate the Efficacy of BAY 43-9006 (Sorafenib) in Metastatic Renal Cell Carcinoma
Brief Title: Sorafenib in Treating Patients Who Are Undergoing Surgery for Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02920; NCI-2012-02920 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000438709; 2004-0516 (Other: M D Anderson Cancer Center); 6630 (Other: CTEP); P30CA016672 (NIH); N01CM62202 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

ARMS (3):
- Group I (cytoreductive nephrectomy and sorafenib tosylate) (Experimental): Patients undergo cytoreductive nephrectomy on day 1. Patients then receive oral sorafenib twice daily on days 15-84.
  In all groups, patients with stable or regressing disease continue to receive oral sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Some patients may continue treatment for longer than 1 year at the discretion of the investigator.
  Interventions: Procedure: therapeutic conventional surgery; Drug: sorafenib tosylate; Other: laboratory biomarker analysis
- Group II (sorafenib tosylate and cytoreductive nephrectomy) (Experimental): Patients receive oral sorafenib twice daily on days 1-7. Patients undergo cytoreductive nephrectomy on day 8. Patients then receive oral sorafenib twice daily on days 22-84.
  In all groups, patients with stable or regressing disease continue to receive oral sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Some patients may continue treatment for longer than 1 year at the discretion of the investigator.
  Interventions: Procedure: therapeutic conventional surgery; Drug: sorafenib tosylate; Other: laboratory biomarker analysis
- Group III (sorafenib tosylate and cytoreductive nephrectomy) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Patients undergo cytoreductive nephrectomy on day 29. Patients then receive oral sorafenib twice daily on days 43-84.
  In all groups, patients with stable or regressing disease continue to receive oral sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Some patients may continue treatment for longer than 1 year at the discretion of the investigator.
  Interventions: Procedure: therapeutic conventional surgery; Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo cytoreductive nephrectomy
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sorafenib before and after surgery may be an effective treatment for kidney cancer. This phase II trial is studying how well sorafenib works in treating patients who are undergoing surgery for metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Efficacy of BAY 43-9006 (sorafenib tosylate) by evaluating response rate. II. Toxicities of BAY 43-9006 in metastatic renal cell carcinoma (RCC). III. Intraoperative and peri/postoperative safety of BAY 43-9006.

SECONDARY OBJECTIVES:

I. Time to progression. II. Duration of response. II. Overall Survival.

TERTIARY OBJECTIVES:

I. Tissue expression of VEGFR-2/phospho-VEGFR-2, PDGFR/phospho-PDGFR, FGFR/phospho-FGFR, ERK/phospho-ERK, RAF-1/phospho-RAF-1, p38/phospho-p38, Akt/phospho-Akt, P27, Ki67, TGF-alpha, and TUNEL pre- and post- therapy (optional studies).

II. Oligonucleotide analysis of tissue pre- and post-therapy (optional studies).

OUTLINE: This is a non-randomized study. Patients are sequentially assigned to 1 of 3 treatment groups.

GROUP I: Patients undergo cytoreductive nephrectomy on day 1. Patients then receive oral sorafenib twice daily on days 15-84.

GROUP II: Patients receive oral sorafenib twice daily on days 1-7. Patients undergo cytoreductive nephrectomy on day 8. Patients then receive oral sorafenib twice daily on days 22-84.

GROUP III: Patients receive oral sorafenib twice daily on days 1-28. Patients undergo cytoreductive nephrectomy on day 29. Patients then receive oral sorafenib twice daily on days 43-84.

In all groups, patients with stable or regressing disease continue to receive oral sorafenib twice daily for up to 1 year in the absence of disease progression or unacceptable toxicity. Some patients may continue treatment for longer than 1 year at the discretion of the investigator.

After completion of study treatment, patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 45 patients (15 per treatment group) will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic clear cell RCC who are eligible for cytoreductive nephrectomy as agreed upon by Medical Oncology and Urology team members; patients with metastatic disease eligible for cytoreductive nephrectomy should have the following characteristics: resectable primary tumor (no gross adjacent organ invasion, no or minimal abdominal lymphadenopathy, no or minimal inferior vena caval involvement), bulk of metastatic disease within the primary tumor, absence of multiple liver metastases, no more than 2 organ sites involved with metastases
* Patients must have measurable disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >= 20 mm with conventional techniques or >= 10 mm with spiral computed tomography (CT) scan
* ECOG performance status =< 1
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hgb > 9.0 g/dL
* Total bilirubin =< 2.0 mg/dl
* Albumin > 3.0 g/dL
* Serum creatinine =< 2.0 mg/dl
* AST (SGOT) and/or ALT (SGPT) =< 2.5 x institutional upper limit of normal for subjects without evidence of liver metastases
* AST (SGOT) and/or ALT (SGPT) =< 5 X institutional upper limit of normal for subjects with documented liver metastases
* Female patients of childbearing potential must have a normal plasma beta human chorionic gonadotropin (beta-HCG) within 24 hours prior to enrolling in the study due to the possible teratogenic effect; however, patients will be eligible if their beta-HCG is elevated and is determined to be due to malignancy
* Patients of child fathering or childbearing potential must agree to practice a form of medically acceptable birth control while on study
* Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution; patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy
* Patients must have ability to comply with study and/or follow-up procedures
* Prior biopsy material (blocks or unstained slides) must be available for comparison purposes

Exclusion Criteria:

* No prior malignancy is allowed, except for non-melanoma skin cancer, in situ carcinoma of any site, or other cancers for which the patient has been adequately treated and disease free for 5 years
* Patients must not have received any systemic anticancer therapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients must not be scheduled to receive another experimental drug while on this study; patients are permitted to be on concomitant bisphosphonates
* Patients who are incapable of swallowing pills are excluded from this study
* Patients must not have a primary brain tumor, any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of stroke
* Patients must not have active acute infections that could be worsened by anticancer therapy or interfere with this study
* Patients must not have clinically significant cardiovascular disease, recent myocardial infarction (i.e. last 6 months), (unstable angina), New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac dysrhythmia requiring medication, or peripheral vascular disease (grade II or greater)
* Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Patients with uncontrolled hypertension > 140/90 are excluded from the study
* Patients must not have any history of bleeding diathesis; patients must not be on therapeutic anticoagulation; prophylactic anticoagulation (i.e. low dose coumadin) of venous or arterial access devices is allowed provided that the requirements for PT, INR or PTT are met
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with BAY 43-9006
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 11, 2006 to July 12, 2007. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: This trial was run at the same time as a competing trial and suffered from poor accrual. For that reason it was closed.
Groups:
- Cytoreductive Nephrectomy Day 0: Group 1: Immediate cytoreductive nephrectomy, two weeks rest, and 10 weeks Sorafenib 400 mg orally mouth twice a day.
- Sorafenib + Cytoreductive Nephrectomy Day 8: Group 2: One week Sorafenib 400 mg orally mouth twice a day, cytoreductive nephrectomy, two weeks rest, 9 weeks Sorafenib
- Sorafenib + Cytoreductive Nephrectomy Day 29: Group 3: Four weeks Sorafenib 400 mg orally mouth twice a day, Cytoreductive Nephrectomy, two weeks rest, 6 weeks Sorafenib
Period: Overall Study
Arm/Group | Cytoreductive Nephrectomy Day 0 | Sorafenib + Cytoreductive Nephrectomy Day 8 | Sorafenib + Cytoreductive Nephrectomy Day 29
Started | 3 | 3 | 4
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cytoreductive Nephrectomy Day 0 | Sorafenib + Cytoreductive Nephrectomy Day 8 | Sorafenib + Cytoreductive Nephrectomy Day 29 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 2 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of BAY 43-9006 by Evaluating Response Rate
Description: Response rate (participants with response/total number participants) where number of participants with response evaluated using international criteria proposed by (RECIST) Committee of: Complete Response: Disappearance all target lesions; Partial Response (PR): > 30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD. Progressive Disease (PD): > 20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance of 1 or > new lesions; Stable Disease:
  Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started.
Time Frame: Every 2 weeks during 4 week cycle
Population: Unable to assess response due to small sample size.
Arm/Group | Cytoreductive Nephrectomy Day 0 | Sorafenib + Cytoreductive Nephrectomy Day 8 | Sorafenib + Cytoreductive Nephrectomy Day 29
Number analyzed (Participants) | 0 | 0 | 0

2. Other Pre Specified Outcome: Duration of Overall Response
Description: Duration of overall response is measured from the time measurement criteria are met for Complete Response or Partial Response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started), measured in days.
Time Frame: Following 10 weeks of treatment, followed every 2 weeks or until disease progression
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Overall Survival
Description: The number of participants surviving from baseline (treatment) to death due to any cause measured in days.
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Time to Progression
Description: Time, in weeks, after treatment until disease progresses. Repeat radiologic studies to evaluate disease progression or response after 10 weeks of BAY 43 9006 therapy.
Time Frame: Following 10 weeks of treatment or until disease progression
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Groups:
- Sorafenib + Cytoreductive Nephrectomy: All participants received Sorafenib 400 mg orally mouth twice a day for a total of 10 weeks over the course of the study and had surgical procedure Cytoreductive Nephrectomy before treatment with Sorafenib or in between courses of Sorafenib
Arm/Group | Sorafenib + Cytoreductive Nephrectomy
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Cytoreductive Nephrectomy (N=10)
hyperuricemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Cytoreductive Nephrectomy (N=10)
alopecia (General disorders) | 2
anorexia (Gastrointestinal disorders) | 1
cough (General disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 1
diarrhea (Gastrointestinal disorders) | 4
dizziness (General disorders) | 1
dysphagia (Gastrointestinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
edema:head and neck (General disorders) | 1
fatigue (General disorders) | 10
hand foot syndrome (Skin and subcutaneous tissue disorders) | 1
hematoma (General disorders) | 1
hemoglobin (Blood and lymphatic system disorders) | 4
hemoglobinuria (Blood and lymphatic system disorders) | 1
hypertension (Blood and lymphatic system disorders) | 2
hyperuricemia (Blood and lymphatic system disorders) | 1
hypoalbuminemia (Blood and lymphatic system disorders) | 1
hypomagnesemia (Blood and lymphatic system disorders) | 4
hyponatremia (General disorders) | 1
hypophosphatemia (Blood and lymphatic system disorders) | 2
infection (other), (Infections and infestations) | 1
leukocytes (Blood and lymphatic system disorders) | 2
lymphopenia (Blood and lymphatic system disorders) | 1
mucositis (General disorders) | 4
nausea (Gastrointestinal disorders) | 3
neutrophils (ANC) (Blood and lymphatic system disorders) | 1 — ANC = Absolute Neutrophil Count
pain (chest/thorax) (Investigations) | 1
pain (joint) (Musculoskeletal and connective tissue disorders) | 1
platelets (Blood and lymphatic system disorders) | 3
proteinuria (Renal and urinary disorders) | 1
rash/desquamation (Skin and subcutaneous tissue disorders) | 4
secondary malignancy (Investigations) | 1
vomiting (Gastrointestinal disorders) | 1
watery eye (Eye disorders) | 1
weight loss (Gastrointestinal disorders) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Study ended early due to early termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less